CLINICAL TRIAL: NCT06638697
Title: CREM - Reference Center for Aging and Movement: Clinical and Functional Outcomes in a Controlled Clinical Trial with Older Adults
Brief Title: CREM - Clinical and Functional Outcomes in a Controlled Clinical Trial with Older Adults
Acronym: CREM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Andrea Kruger Goncalves, Doctor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 36044620.5.0000.5336
Record Dates: First submitted 2024-10-02; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Aged; Aged Subject
Keywords: elderly; functionality; physical exercise; cognition; physical fragility; physical fitness
MeSH Terms: conditions — Motor Activity | interventions — Nordic Walking; Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- exercise program (Experimental): Participants will receive intervention of different physical training for 32 weeks and will be periodized in an equivalent way.
  Interventions: Other: Free walking; Other: Nordic walking; Other: Dance; Other: Physical exercise for cognition; Other: Balance; Other: Aquatic physiotherapy; Other: Multicomponent gymnastics; Other: Water aerobics; Other: Hydroposture; Other: deep water walking; Other: Weight training; Other: Mat pilates

INTERVENTIONS:
Other: Free walking — The free walking training program will last 32 weeks. The intensity of the training will be controlled by the scale of perceived exertion (Borg). The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial stretching and the final stretching will last five minutes.
Other: Nordic walking — The Nordic walking training program will last 32 weeks. The intensity of the training will be controlled by the Borg scale of perceived exertion. The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial and final stretching will last five minutes.
Other: Dance — The Dance training program will last 32 weeks. The intensity of the training will be controlled by the Borg scale of perceived exertion. The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial and final stretching will last five minutes.
Other: Physical exercise for cognition — The Physical exercise for cognition training program will last 32 weeks. The intensity of the training will be controlled by the Borg scale of perceived exertion. The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial and final stretching will last five minutes.
Other: Balance — The Balance training program will last 32 weeks. The intensity of the training will be controlled by the Borg scale of perceived exertion. The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial and final stretching will last five minutes.
Other: Aquatic physiotherapy — The Aquatic Physiotherapy training program will last 32 weeks. The intensity of the training will be controlled by the Borg scale of perceived exertion. The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial stretching and the final stretching will last five minutes.
Other: Multicomponent gymnastics — The Multicomponent Gymnastics training program will last 32 weeks. The intensity of the training will be controlled by the Borg scale of perceived exertion. The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial stretching and the final stretching will last five minutes.
Other: Water aerobics — The Water Aerobics training program will last 32 weeks. The intensity of the training will be controlled by the Borg scale of perceived exertion. The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial stretching and the final stretching will last five minutes.
Other: Hydroposture — The Hydroposture training program will last 32 weeks. The intensity of the training will be controlled by the Borg scale of perceived exertion. The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial stretching and the final stretching will last five minutes.
Other: deep water walking — The deep water walking training program will last 32 weeks. The intensity of the training will be controlled by the Borg scale of perceived exertion. The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial stretching and the final stretching will last five minutes.
Other: Weight training — The weight training program will last 32 weeks. The intensity of the training will be controlled by the Borg scale of perceived exertion. The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial stretching and the final stretching will last five minutes.
Other: Mat pilates — The MAt pilates program will last 32 weeks. The intensity of the training will be controlled by the Borg scale of perceived exertion. The training program will have a frequency of two sessions per week, lasting 60 minutes and will be divided into three parts: a) stretching, joint mobility and warm-up; b) main part (according to the objectives of each modality); c) cool-down and final stretching. Both the initial stretching and the final stretching will last five minutes.

SUMMARY:
To evaluate and compare the effects of different types of physical exercise on clinical and functional outcomes in the elderly. 240 community-dwelling elderly individuals of both sexes, sedentary, will be recruited for twelve groups of elderly individuals who will receive intervention for 32 weeks of different types of physical exercise (free walking, Nordic walking, dancing, physical exercise for cognition, balance, aquatic physiotherapy, multicomponent gymnastics, water aerobics, hydro-postural exercises, aquatic jogging, weight training, and Pilates mat). The training programs will have a frequency of two sessions per week and will last 50 minutes and will be periodized so that the duration of the sessions is equal among them. In order to evaluate the effects of the training, evaluations will be carried out before, during and after the training period of functional fitness, clinical-functional and biomechanical parameters. It is expected that the intervention groups will present results according to the nature of the modality and that they will be more effective when compared to the control group. As well as improvements in the variables of gait speed, muscle strength, balance and cognition.

ELIGIBILITY:
Inclusion Criteria:

* elderly people over 60 years old,
* sex female our male,
* presenting medical authorization to practice exercises,
* being able to understand verbal instructions for carrying out the tests,
* having accessibility to carry out the training,
* coming from local Health Units and the community,
* presenting independent walking and not having participated in any physical activity for at least three months before starting the research.

Exclusion Criteria:

* not having a medical certificate indicating that they are fit to perform physical activity,
* presenting medical comorbidities and/or a medical condition that contraindicates participation in the study, severe heart disease, uncontrolled arterial hypertension, myocardial infarction within a period of less than one year or history of physical-cognitive impairment, sequelae of a stroke,
* having a pacemaker,
* having undergone recent surgery,
* prosthetics in the lower limbs or neuropathic pain in the lower limbs.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Lower Limb Strength | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  Five-Repetition Sit-to-Stand Test - This assesses the time it takes for an individual to stand up so that their knees are fully extended and then sit down again as quickly as possible. Individuals with 5-repetition times for this test greater than the following may be considered to have poorer than average performance: 11.4 sec (60 to 69 years), 12.6 sec (70 to 79 years), and 14.8 sec (80 to 89 years).
Upper limb strength | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  Dynamometry - Obtained using a hand-held dynamometer. The subject is seated and asked to exert as much force as possible with the dominant upper limb. The highest strength value obtained will be considered, adjusted by the body mass index (in quartiles) and stratified by sex.
Upper limb flexibility | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  Reach Behind the Back - While standing, the subject places the preferred hand on the same shoulder, palm open and fingers extended, reaching as far as possible toward the middle of the back. The hand of the other arm is placed behind the back, palm up, reaching as far as possible, in an attempt to touch or overlap the extended middle fingers of the other hand. Measured in distance (cm).
Lower limb flexibility | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  Sitting and Reaching - The subject remains seated in the chair and with one leg extended, tries to reach the toes, it is measured in distance (cm).
Aerobic endurance | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  6-Minute Walk Test - On a 30-meter course, participants walk as fast as possible (without running) around the course as many times as they can within the time limit, it is measured in distance (m) and reflects aerobic endurance
Static balance | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  Single-leg support tests - Static balance tests (Single-leg 30 seconds). The ability of subjects to stand on the force platform in a single-leg position with their eyes open. The position is standing on one foot (single-leg support), the subject chooses whether the right or left leg, looking at a fixed point in line with the eyes. The task is timed until the subjects return the foot to the ground or reach the maximum time of 30 seconds. The force platform will be used and the rate of displacement of the COP will be analyzed in the anteroposterior (Fx), mediolateral (Fy) and vertical (Fz) axes.
Dynamic balance | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  Timed and Up and Go (TUG) - The patient starts by sitting in a chair, walks a distance of 3 meters, goes around a cone (180º turn), returns and sits back down in the chair. The patient is instructed to perform the test as quickly as possible. For classification: test performed in up to 10 seconds (healthy elderly, independent and without risk of falls); test between 11 and 20 seconds (frail elderly, with partial independence and low risk of falls); time greater than 20 seconds (significant deficit in physical capacity, high risk of falls and dependence in ADLs).
Walking speed | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  Ten-meter walk test - The ten-meter walk test will be used to assess self-selected walking speed (VAS). The time taken to walk ten meters will be recorded. The individual will be given the following command: "I want you to walk at a comfortable speed, the one that is most similar to your daily pace. The average time of three attempts will be used to calculate the walking speed expressed in meters per second (m/s).

SECONDARY OUTCOMES:
Concern about falls | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  Falls Efficacy Scale International (FES-I) - The FES-I is a scale for assessing self-efficacy related to falls. The instrument presents questions about concern about the possibility of falling when performing 16 activities, with respective scores from one to four. The total score can range from 16 points (no concern) to 64 points (extreme concern).
Pain index | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  McGill Pain Questionnaire - The instrument is used to measure the quality and intensity of pain, the patient chooses between 15 words and the pain is classified in its sensory and affective dimensions, along with an analog scale that evaluates the general intensity of pain in the last few days and a 6-item scale with a global description of intensity.
Depressive symptoms | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  Geriatric Depressive Symptoms (GDS-15) - The GDS-15 is a widely used and validated scale as a diagnostic instrument for depression in the elderly. It is a self-assessed scale for assessing depressive symptoms, consisting of 15 questions, in which a score of five or more points is indicative of a probable depressive episode.
Cognition | Assessments will take place before, during and after the training period at three times: 1) Pre-intervention (0 weeks), 2) after 16 weeks of training, 3) Post-intervention (32 weeks).
  General cognition - evaluated with the Montreal Cognitive Assessment (MoCA). It covers various cognitive domains (visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall, and orientation). Scores on the MoCA can range from 0 to 30, with higher scores indicating better cognitive function. Participants will be classified in cognitively unimpaired (CU), mild cognitive impairment (MCI), and dementia according to the total MoCA score.

IPD SHARING:
Plan to Share IPD: No